CLINICAL TRIAL: NCT06353451
Title: Smartphone Screen Time Reduction Improves Mental Health: A Randomized Clinical Trial
Brief Title: Digital Detox Study: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danube University Krems (Other)
Responsible Party: Principal Investigator, Christoph Pieh, Full Professor and Head of Department, Danube University Krems
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EK GZ 67/2021-2024
Record Dates: First submitted 2024-03-19; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-03

CONDITIONS: Health Behavior
Keywords: Smartphone screen time; Digital Detox; Social Media Detox
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: Two groups, non blinded, randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Smartphone screen time should be reduced to less than 2 hours per day for 3 consecutive weeks. Screen time will be controlled by screenshots weekly.
  Interventions: Behavioral: Digital Detox
- Control group (No Intervention): Smartphone usage behavior should continue unchanged. Screen time will be measured by uploaded screenshots weekly.

INTERVENTIONS:
Behavioral: Digital Detox — In the intervention group, smartphone screen time will be reduced to less than 2 hours for 3 consecutive weeks.
  Arms: Intervention Group

SUMMARY:
The aim of the present RCT is to investigate the effect of smartphone screen time reduction on mental health indicators in healthy, 18-29 yo Austrian students.

After inclusion and randomization to intervention- and control group, normal screen time behavior will be assessed for 10-days. After that, the mental health parameters will be carried out in both groups as a baseline survey (T0). After that, intervention group should limit smartphone screen time to less than 2 hours per day for three consecutive weeks. Control group should use smartphones as usual. After that, mental health parameters will be assessed again in both groups (post-intervention, T1). After T1, there are no further requirements regarding screen time. Mental health parameters will be assessed again in both groups at follow-up (T2).

Main outcome parameters are 1) Well-Being (WHO-5), depressive symptoms (PHQ-9), stress (PSQ-20), and sleep quality (ISI).

The primary hypothesis (stated at Open Science Framework before Enrollment: https://osf.io/a9k76) is that mental health indicators, particularly stress, depressive symptoms, and sleep quality will improve throughout the intervention compared to the control group as well as to baseline.

DETAILED DESCRIPTION:
According to the power-analysis (small to medium effect size of d=.45, power .8, significance level < .05, icc = .05), a sample of N > 100 should be recruited through newsletter, notices and social media. The inclusion criteria are more than 3 hours of screen time per day, no mental disorder, no ongoing psychotherapy or use of psychotropic drugs.

After signing the informed consent, participants have to download an App (ESMira®), which processes the whole study. The first step is to fill out sociodemographic data, smartphone use and mental health questionnaires. After controlling for inclusion- and exclusion criteria, ESMira will randomize into intervention- (IG) and control group (CG). Participants in the control group (CG) should continue their smartphone behavior unchanged throughout the entire study period. Participants in the intervention group (IG) should continue their smartphone usage unchanged for the first 10 days (Baseline.) After that, the mental health parameters will be carried out in both groups as a baseline survey (T0). After that, participants of the intervention group should limit their smartphone screen time under two hours per day for three weeks. To comply with that, participants should use the limiter function of their smartphone or download an additional app. A screen shot of the screen time has to be uploaded weekly on Monday for the previous week (Monday to Sunday). At the end of the intervention (t1), the mental health questionnaires will be collected again in both groups. After T1, there are no further requirements regarding screen time. Mental health parameters will be assessed again in both groups at follow-up (T2).

During the study period participants will be asked to additionally wear a fitness tracker to measure daily movement as well as objective stress parameters.

Data collection and randomization The whole data collection procedure will be carried out through the ESMira App. ESMira is a tool for running longitudinal studies (ESM, AA, EMA, ...) with completely anonymized communication with participants and data collection.

Smartphone screen time Weekly screen time will be documented in both groups using the smartphones' built-in screen time measurements.

Statistical plan

Repeated measurements ANOVAs (rm-ANOVA) will be applied to analyze differences. Difference between t0 (baseline) and t1 (post-intervention) in the intervention group and on the difference between control group and intervention group are the primary hypotheses. Effects (between- as well as within group) will be analyzed for all 3 measurement points as well. Furthermore, a secondary analysis will be applied to analyze the sub-sample that strictly adhered to the time limits.

In case of baseline group-differences, variables will be added as covariates in the rm-ANOVA. A Greenhouse-Geisser correction will be applied, if sphericity assumption is violated. In the post hoc tests, Bonferroni correction will be applied to adjust for multiple comparisons.

Missing values will be dealt with via maximum likelihood estimation. Percentage changes in the main outcomes between baseline and post-intervention will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* 18-29 years old
* male/female
* daily screen time > 3 h/d
* no mental disorder
* no ongoing psychotherapy
* no psychotropic drugs

Exclusion Criteria:

* < 18 yo or > 29 yo
* daily screen time < 3 h/d
* mental disorder (self-statement)
* in ongoing psychotherapy
* psychotropic drug use

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-01-21 (Actual); Study Completion 2024-01-21 (Actual)

PRIMARY OUTCOMES:
Depressive Symptoms | The questionnaire will be assessed at 3 time points, 1) at baseline (=immediately pre-intervention (t0), 2) immediatly after the 3-week intervention (t1), and 3) at Follow-Up (t2= six weeks post intervention).
  Patient Health Questionnaire (PHQ-9):
  The PHQ-9 contains nine self-rating items on a four-point scale ranging from 0 ("not at all") to 3 ("nearly every day"), resulting in a total score from 0 to 27. Higher scores indicate more depressive symptoms.
Stress | The questionnaire will be assessed at 3 time points, 1) at baseline (=immediately pre-intervention (t0), 2) immediatly after the 3-week intervention (t1), and 3) at Follow-Up (t2= six weeks post intervention).
  Perceived Stress Questionnaire (PSQ-20):
  Each item is rated from almost never (=1) to usually (= 4), with a sum score from 20 to 80. Higher scores indicate more stress.
Sleep Quality | The questionnaire will be assessed at 3 time points, 1) at baseline (=immediately pre-intervention (t0), 2) immediatly after the 3-week intervention (t1), and 3) at Follow-Up (t2= six weeks post intervention).
  Insomnia Severity Index (ISI):
  The ISI comprises 7 self-reported items, each rated on a scale from 0 to 4, resulting in sum scores from 0 to 28. Higher scores indicate more insomnia symptoms or less sleep quality.
Well-being | The questionnaire will be assessed at 3 time points, 1) at baseline (=immediately pre-intervention (t0), 2) immediatly after the 3-week intervention (t1), and 3) at Follow-Up (t2= six weeks post intervention).
  World Health Organization well-being questionnaire (WHO-5):
  The WHO-5 contains 5 items (0 to 5 points). Scores range from 0 (no well-being) to 25 points (maximal well-being).

SECONDARY OUTCOMES:
Problematic smartphone use | The questionnaire will be assessed at 3 time points, 1) at baseline (=immediately pre-intervention (t0), 2) immediatly after the 3-week intervention (t1), and 3) at Follow-Up (t2= six weeks post intervention).
  Smartphone Addiction Scale Short Version (SAS-SV):
  The 10 items range from 1 (=strongly disagree) to 6 (=strongly agree) points with a sum score from 10 to 60. Higher scores indicate problematic smartphone use.
Body Appreciation | The questionnaire will be assessed at 3 time points, 1) at baseline (=immediately pre-intervention (t0), 2) immediatly after the 3-week intervention (t1), and 3) at Follow-Up (t2= six weeks post intervention).
  Body Appreciation Scale-2 (BAS-2):
  The scale is comprised of 10 items, which can be rated from "never" (1) to "always" (5). Higher scores indicate a more positive body appreciation.
Anxiety Symptoms | The questionnaire will be assessed at 3 time points, 1) at baseline (=immediately pre-intervention (t0), 2) immediatly after the 3-week intervention (t1), and 3) at Follow-Up (t2= six weeks post intervention).
  Generalized Anxiety Disorder 7 scale (GAD-7):
  The GAD-7 contains 7 self-rating items on a four-point scale, from 0 to 3 (maximum score 21). Higher scores indicate more anxiety symptoms.
Eating Disorder | The questionnaire will be assessed at 3 time points, 1) at baseline (=immediately pre-intervention (t0), 2) immediatly after the 3-week intervention (t1), and 3) at Follow-Up (t2= six weeks post intervention).
  SCOFF (Sick, Controll, One stone, Fat, Food) Questionnaire:
  Five items can be answered with "yes"=1 or "no"=0. The total score ranges from 0 to 5. A total score of 2 or above indicates disordered eating.

OTHER OUTCOMES:
Physical Activity | Physical activity was recorded from the beginning of the baseline phase for the duration of 5 weeks (2 weeks baseline, 3 weeks intervention) and stopped after intervention (=t1).
  Physical activity (moderate to high intensity physical activity in minutes per day) was assessed with a Fitness Tracker (Fitbit® Inspire 3).
Heart rate variability (HRV) | HRV was recorded from the beginning of the baseline phase for the duration of 5 weeks (= 2 weeks baseline, 3 weeks intervention) and stopped after intervention (=t1).
  HRV was measured regularly every day and then an overall score was created for the sleep period using a Fitness Tracker (Fitbit® Inspire 3).
Resting Heart Rate (RHR) | RHR was recorded from the beginning of the baseline phase for the duration of 5 weeks (= 2 weeks baseline, 3 weeks intervention) and stopped after intervention (=t1).
  RHR was measured regularly every day and then an overall score was created for the sleep period using a Fitness Tracker (Fitbit® Inspire 3).
Screen time | Starting with the baseline screening (November 10th, 2023) weekly until Follow-Up (t2=January 21st, 2024)
  Smartphone screen time will be assessed weekly from November 10th, 20223 until January 21st, 2024 using the smartphones' built-in screen time measurements. Every Monday, participants will received a push-up message via the ESMira app to upload the screenshot from their screen time of the previous week (Monday to Sunday), including the amount spent on social media sites. If necessary, participants received up to three reminders.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Pieh, MD, Principal Investigator — Danube University Krems
Locations (1):
- Danube University Krems, Krems, Lower Austria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dale R, Haider K, Majdandzic J, Hoenigl A, Schwab J, Pieh C. The influence of smartphone reduction on heart rate variability: a secondary analysis from a randomised controlled trial. Health Psychol Behav Med. 2025 Aug 16;13(1):2546376. doi: 10.1080/21642850.2025.2546376. eCollection 2025. PMID 40831581

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-08): https://cdn.clinicaltrials.gov/large-docs/51/NCT06353451/Prot_SAP_000.pdf